CLINICAL TRIAL: NCT05638347
Title: Use the Protocol Title. A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and the Food Effect on the Pharmacokinetics of HRS-7085 in Healthy Participants
Brief Title: A Trial of HRS-7085 Tablet in Healthy Participants With and Without Food Effect.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HRS-7085-102-AUS
Record Dates: First submitted 2022-11-27; First posted 2022-12-06 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Part 1: HRS-7085 Single Ascending Dose (SAD) Both males and females are planned to be enrolled in five cohorts (optional and determined by Safety Review Committee (SRC) in this SAD study Part 2: Food Effect: Participants in cohort 3 who have finished the follow-up visit will be involved in the food effect study after safety evaluation by the investigator.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-7085 tablets Cohort 1 (Experimental): Part 1- HRS-7085 tablets
  Interventions: Drug: HRS-7085 tablets; Drug: Placebo tablet
- HRS-7085 tablets Cohort 6 (Experimental): Part 1- HRS-7085 tablets
  Interventions: Drug: HRS-7085 tablets; Drug: Placebo tablet

INTERVENTIONS:
Drug: HRS-7085 tablets — Single oral administration
Drug: Placebo tablet — Single oral administration

SUMMARY:
The study is being conducted to evaluate the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of HRS-7085.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, volunteers to participate in the trial.
2. Male or female aged between 18 years and 55 years (inclusive) at the date of signed consent form.
3. Total body weight 45 kg~100 kg (inclusive) at screening, and body mass index (BMI) between 18 and 32 kg/m2 (inclusive).
4. For healthy subjects, no clinically significant abnormalities.
5. Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods

Exclusion Criteria:

1. Known medical history of severe disease in cardiovascular, liver, kidney, digestive tract, mental nerve, hematology, metabolic disorders, etc.
2. Severe injuries or major surgeries within 3 months before dosing.
3. Subjects with infectious disease.
4. Live/attenuated vaccine within 3 months prior to dosing or any vaccine during the trial.
5. Blood donation or loss of ≥ 200 mL of blood within 1 month prior to dosing, or ≥ 400 mL of blood within 3 months prior to dosing; or receive a blood transfusion within 2 months prior to dosing.
6. Clinically significant abnormalities in 12-Lead ECG
7. More than 5 cigarettes daily (or products with equivalent amount of nicotine) for 3 months prior to screening, or positive cotinine test at screening or baseline.
8. Positive urine drug at screening or baseline.
9. Subject who cannot perform venous blood sampling.
10. Known history or suspected of being allergic to the study drugs and their excipients.
11. Use of prescription medicine within 2 weeks, or OTC medicine, within 1-week or 5 half-lives prior to dosing.
12. History of alcohol abuse within 3 months prior to screening, or positive alcohol breath test at screening or baseline.
13. Participation in clinical trials of other investigational drugs or medical devices within 1 month or 5 half-lives prior to dosing.
14. Special dietary requirements that cannot follow the meal plan in the food effect study.
15. In the investigator's judgment, may increase the risk to the subject.
16. Unwilling or unable to comply with the Lifestyle Guidelines detailed in this protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Start of Treatment to end of study approximately 1 week

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 1 week)
  Area under the concentration-time curve from time 0 to last time point after HRS-7085 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 1 week)
  Area under the concentration-time curve from time 0 to infinity after HRS-7085 administration
Pharmacokinetics-Tmax | Start of Treatment to end of study (approximately 1 week)
  Time to Cmax of HRS-7085
Pharmacokinetics-Cmax | Time Frame: Start of Treatment to end of study (approximately 1 week)
  Maximum observed concentration of HRS-7085
Pharmacokinetics-CL/F | Time Frame: Start of Treatment to end of study (approximately 1 week)
  Apparent clearance of HRS-7085
Pharmacokinetics-Vz/F | Time Frame: Start of Treatment to end of study (approximately 1 week)
  Apparent volume of distribution during terminal phase of HRS-7085
Pharmacokinetics-t1/2 | Time Frame: Start of Treatment to end of study (approximately 1 week)
  Terminal elimination half-life of HRS-7085

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia